CLINICAL TRIAL: NCT03092778
Title: Percutaneous Image Guided Cryoablation of the Vagus Nerve for Management of Mild-Moderate Obesity
Brief Title: Cryoablation for Obesity Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Endocare, Inc. (Industry)
Responsible Party: Principal Investigator, John Prologo, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00095192
Record Dates: First submitted 2017-03-24; First posted 2017-03-28 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Obesity
Keywords: Cryoablation; Radiology
MeSH Terms: conditions — Obesity | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cryoablation Group (Experimental): Participants with mild to moderate obesity will undergo a cryoablation procedure to the vagal nerve.
  Interventions: Procedure: Cryoablation

INTERVENTIONS:
Procedure: Cryoablation — A computed tomography (CT) scan will be completed to map out where to insert the cryoablation needle. Numbing medicine will be used to numb the skin and deeper tissues before inserting the needle.
  The cryoablation needle will be inserted and directed toward the target area of the vagal nerve. A CT scan will be done during the procedure to help guide the needle which will be held in position by the study doctor(s) once it reaches the target area. With the needle in place, the study doctor(s) will freeze the zone over 3 minutes, a 2 minutes thaw will follow, then 2 more cycles of 3 minutes freeze and 2 minute thaw will complete the procedure. This portion of the procedure can last from 25 to 35 minutes. Once the targeted area has been properly treated, the cryoablation needle will be withdrawn.

SUMMARY:
The purpose of this study is to assess the efficacy of cryoablation therapy for the treatment of mild to moderate obesity and test the safety (good and bad effects) of this procedure. The vagus nerve transmits hunger signals from the stomach to the brain, and in response transmits stomach expansion signals from the brain to the stomach. Investigators believe that by interrupting this communication, participants could experience less hunger and in turn lose weight.

DETAILED DESCRIPTION:
The purpose of this single arm study is to assess the efficacy of cryoablation therapy for the treatment of mild to moderate obesity and test the safety (good and bad effects) of this procedure. The vagus nerve transmits hunger signals from the stomach to the brain, and in response transmits stomach expansion signals from the brain to the stomach.Investigators believe that by interrupting this communication, participants could experience less hunger and in turn lose weight.

The rationale for using cryoablation to treat obesity is based on this investigator's experience safely targeting peripheral nerves via CT guidance and treated with thermal ablation in daily clinical practice. the primary objective of this research is to evaluate the feasibility and safety (over time) of percutaneous image guided cryoablation of the posterior vagus nerve in obese patients. The secondary objective consist of temporal evaluation of weight loss and appetite before and after the procedure. This will be analyzed through documentation of weight, and through the implementation of validated outcome instruments.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 30-35
* Weight loss refractory to diet changes or exercise
* Absence of coagulopathy
* Ability and willingness of patient to provide written informed consent

Exclusion Criteria:

* Active infection
* Underlying congenital anatomic or other spinal anomalies that result in non-conventional anatomy at the gastro-esophageal junction
* Pregnant or planning to become pregnant
* Immunosuppression
* History or laboratory results indicative of any significant cardiac, endocrine, hematologic, hepatic, immunologic, infectious, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric, renal, neoplastic, or other disorder that in the opinion of the Principal Investigator would preclude the safe performance of cryoablation
* Uncorrectable coagulopathies
* Concurrent participation in another investigational trial involving systemic administration of agents or within the previous 30 days
* Have undergone a previous bariatric surgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
Number of Cryoablation Procedure Events (CPEs) | Post Intervention (Up to 24 Hours)
  Adverse events which occur within the first 24 hours following cryoablation.
Number of Adverse Events | Duration of Study (Up to 2 Years)
  Clinical signs or symptoms of infection (fever), hemorrhage (pain, imaging changes), that occur outside of the time periods specified for CPEs.
Number of Significant Adverse Events (SAEs) | Duration of Study (Up to 2 Years)
  Significant adverse events include life-threatening adverse events and death.
Number of Breakthrough Events | Duration of Study (Up to 2 Years)
  The number of events requiring emergency or urgent physician consultation.
Frequency of Breakthrough Events | Duration of Study (Up to 2 Years)
  The frequency of events requiring emergency or urgent physician consultation.

SECONDARY OUTCOMES:
Weight | Baseline, Month 6 (Post Intervention)
  Weight will be measured in kilograms.
Height | Baseline, Month 6 (Post Intervention)
  Height will be measured in inches.
Body Mass Index (BMI) | Baseline, Month 6 (Post Intervention)
  Body Mass Index will be measured using a BMI calculator.
Hip Circumference | Baseline, Month 6 (Post Intervention)
  Hip Circumference will be measured in inches.
Food Frequency Questionnaire (FFQ) | Week 1, Month 6 (Post Intervention)
  The FFQ is a self-reported measure where participants are asked to describe their food intake during specific time periods.
Kaiser Physical Activity Survey (KPAS) | Week 1, Month 6 (Post Intervention)
  The KPAS is a self-report measure regarding physical activity and living habits. There are four different sections; household and family care activities, occupational activities, active living habits, and participation in sports and exercise. Sections are scored independently on a consecutive scale.
Moorehead-Ardelt Quality of Life Questionnaire | Week 1, Month 6 (Post Intervention)
  The Moorehead-Ardelt Quality of Life Questionnaire is a self-reported measure regarding self-esteem and physical activity levels. Total scores range from -3 to 3, where -3 indicates "very poor" and 3 indicates "very good".
Enrollment Rate | Duration of Study (Up to 2 Years)
  The number of participants enrolled throughout the duration of the study.
Recruitment Rate | Duration of Study (Up to 2 Years)
  The number of participants approached for enrollment throughout the duration of the study.
Retention Rate | Duration of Study (Up to 2 Years)
  The number of participants that complete all study visits.
Exclusion Rate | Duration of Study (Up to 2 Years)
  The number of patients excluded from participation.
Number of Candidates who Chose not to Participate | Duration of Study (Up to 2 Years)
  The number of eligible patients who chose not to participate in the study.
Withdrawal Rate | Duration of Study (Up to 2 Years)
  The number of details regarding patient withdrawal including deaths and lost to followup.
Protocol Deviation Rate | Duration of Study (Up to 2 Years)
  The number of protocol deviations that may impact study results.

CONTACTS AND LOCATIONS:
Overall Officials: David Prologo, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University Hospital, Atlanta, Georgia
  - Emory St. Joseph's Hospital, Atlanta, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia

REFERENCES:
- [Derived] Prologo JD, Lin E, Horesh Bergquist S, Knight J, Matta H, Brummer M, Singh A, Patel Y, Corn D. Percutaneous CT-Guided Cryovagotomy in Patients with Class I or Class II Obesity: A Pilot Trial. Obesity (Silver Spring). 2019 Aug;27(8):1255-1265. doi: 10.1002/oby.22523. PMID 31339003